CLINICAL TRIAL: NCT05411120
Title: Mediterranean-like Unprocessed (CLEAN-MED) Diet Intervention Study of the Gut Microbiome of Healthy Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 10000871; 000871-CC
Record Dates: First submitted 2022-06-04; First posted 2022-06-09 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12-30

CONDITIONS: Diet Therapy
Keywords: Immune System; Gastrointestinal Tract
MeSH Terms: interventions — Diet, Western

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Long-term a Intervention: CLEAN-MED (Experimental): Study arm will consume a Mediterranean like diet, while tracking their food intake for 12 months
  Interventions: Other: CLEAN-MED
- Short-term, Western Diet, high MedDiet score a Intervention: C (Experimental): Study arm will consume a Mediterranean like diet, while tracking their food intake for 9 weeks, With high MEdDIet score.
  Interventions: Other: Western Diet
- Short-term, Western Diet, high MedDiet score a Intervention: W (Experimental): Study arm will consume a Mediterranean like diet, while tracking their food intake for 9 weeks, With high MEdDIet score.
  Interventions: Other: CLEAN-MED
- Short-term, Western Diet, low MedDiet score a Intervention: CL (Experimental): Study arm will consume a western diet eating as they normally would for 9 weeks. With low MEdDIet score.
  Interventions: Other: Western Diet
- Short-term, Western Diet, low MedDiet score a Intervention: We (Experimental): Study arm will consume a Mediterranean like diet, while tracking their food intake for 9 weeks. With low MEdDIet score.
  Interventions: Other: CLEAN-MED

INTERVENTIONS:
Other: Western Diet — Western Diet is by high intakes of pre-packaged foods, refined grains, red meat, processed meat, high-sugar drinks, candy and sweets, fried foods, conventionally-raised animal products, butter and other high-fat dairy products, and low intakes of fruits, vegetables, whole grains.
  Arms: Short-term, Western Diet, high MedDiet score a Intervention: C; Short-term, Western Diet, low MedDiet score a Intervention: CL
Other: CLEAN-MED — Mediterranean like diet is a high consumption of vegetables, oil and moderate consumption of protein, with no processed foods.
  Arms: Long-term a Intervention: CLEAN-MED; Short-term, Western Diet, high MedDiet score a Intervention: W; Short-term, Western Diet, low MedDiet score a Intervention: We

SUMMARY:
Background:

Trillions of tiny organisms-including bacteria, fungi, and viruses-live inside our intestines. These microorganisms break down nutrients in our food, aid our immunity, and help keep us healthy. The population balances among these organisms can vary in different people due to factors including genetics, lifestyle, and diet. More studies are needed to understand how dietary habits affect our intestinal microorganisms.

Objective:

To see how switching from a traditional Western diet (low in fiber, high in saturated fat) to a Mediterranean-like unprocessed foods diet (CLEAN-MED) changes the environment in the intestine. The CLEAN-MED diet includes lots of vegetables, fruits, and whole grains with little sugar or red meat.

Eligibility:

Healthy adults aged 18 to 60

Design:

Participants will be divided into 2 groups. All will start with a trial week. Participants will log all the food they eat and answer questions about their diet throughout the entire study.

Participants in the short-term group will eat a Western diet for 4 weeks and a CLEAN-MED diet for 4 weeks. Food will be provided for the CLEAN-MED diet. Participants will visit the clinic each week and complete surveys. They will log everything they eat. They will provide blood, urine, and stool samples.

Participants in the long-term group will eat the CLEAN-MED diet for up to 12 months. They will visit the clinic each month and complete surveys. They will log everything they eat. They will provide blood, urine, and stool samples. Some foods will be provided for the first 2 weeks. Participants may choose to have a scan of their body composition every few months.

DETAILED DESCRIPTION:
Study Description:

This study (called the CLEAN-MED Diet Study) seeks to examine associations between the gut microbiome, well-being, and adherence to a Mediterranean-like unprocessed food diet. The premise of this study is based on the well-known health benefits of a healthy Mediterranean diet and the potential role that the gut microbiota may serve as a factor in health and disease. The study will recruit healthy outpatient adults, who agree to adhere to a strict Mediterranean-like diet with unprocessed foods, meticulously log their food intake and perceived quality of life using provided questionnaires/tools, and who agree to collect periodic biological samples for analysis. The study will consist of: (1) a short-term cohort who will complete a crossover study design with their habitual Western diet for 4 weeks and the intervention Mediterranean-like unprocessed food diet for 4 weeks (with CLEAN-MED diet food provided by the NIH metabolic kitchen), and (2) a long-term cohort who will continuously adhere to the Mediterranean-like unprocessed food diet for 12 months, following assessment of their baseline diet (with some CLEAN-MED diet foods provided for up to the first 2 weeks of the long-term study, after which the participants must provide their own food).

Objectives:

Primary Objective:

-The primary objective is to measure changes within the gut microbiome in healthy adults who adhere to a Mediterranean-like unprocessed food diet plan.

Secondary Objectives:

* Identify associations between Mediterranean-like unprocessed food diet adherence and psychosocial variables, such as perceived quality of life.
* Identify associations between changes in the gut microbiome and additional biomarkers.

Tertiary Objective:

-Measure the level of adherence to the diet given a strict request for data submission.

Endpoints:

Primary Endpoint:

-Measure changes in gut microbiota composition and functionality from periodic stool sampling using either 16S rRNA and/or shotgun sequencing.

Secondary Endpoints:

* Identify associations between Mediterranean-like unprocessed food diet adherence with perceived quality of life using surveys/questionnaires.
* Measure biomarkers in various biological specimens (stool, blood, and urine) using the pertinent biochemical assays.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Ability of subject to understand and the willingness to sign a written informed consent document
* Age 18-60, at the time of consent
* Willingness to adhere to the dietary regimen and report any major stressors that occur during the study (i.e. changing jobs, moving, death of a close relative/friend, etc.)
* Willingness to provide blood and stool specimens as specified
* BMI >=18 and <= 35 kg/m^2
* Access to necessary resources for participating in a technology-based intervention: computer, smartphone, internet access, etc.
* Has the ability/transportation methods to attend on-site visits
* For 50 of the 60 participants in short-term cohort and for 40 of the 50 participants in the long-term cohort: Currently following a Western diet with PREDIMED-17 MedDiet score <= 7 for >= 1 months and a CLEAN-MED NOVA score of >= 35% kcal in NOVA 4 category with >= 14 items/week in NOVA 4
* For 10 of the 60 participants in short-term cohort and for 10 of the 50 participants in the long-term cohort: Currently following a Western diet with PREDIMED-17 MedDiet score <= 10 for >= 1 months and a CLEAN-MED NOVA score of >= 20% kcal in NOVA 4 category with >= 7 items/week in NOVA 4
* CLEAN-MED Logging Score of >= 43 after initial trial week to continue in the study for the randomization step
* For long-term cohort only: Have resources and capability to consume freshly-cooked (i.e. not pre-packaged or frozen) meals

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study, at the discretion of the PI:

* Current use of medications or dietary supplements for weight or appetite control, whether prescribed or not, including laxatives (within the last 4 weeks)
* Currently eating a vegan, vegetarian, keto or other restrictive diet plan, or food allergies that would affect eating the study diet, at the discretion of the PI
* Active cardiovascular disease (in past year with myocardial infarction, coronary stent or bypass surgery)
* Diabetes (type 1 and 2) or history of gestational diabetes or on hypoglycemic medications or any other indication
* Kidney disease (eGFR less than 50 mL/min per 1.73 m^2)
* Liver disease (liver transaminase higher than 3 times the normal range for the laboratory)
* Symptomatic gallstones
* History of active cancer in the past 3 years except for squamous or basal cell carcinomas of the skin that have been medically managed by local excision
* Has a diagnosed autoimmune condition (i.e. HIV, lupus, etc.) or other immunosuppressive or immunodeficient state, at the discretion of the PI
* Musculoskeletal disorders precluding regular physical activity
* Consumption of the following drugs: proton pump inhibitors, antidiabetic drugs, cholesterol lowering drugs, SGLT-2 inhibitors, GLP-1 receptor agonist, insulin, Amylin analog, Alpha-glucosidase inhibitor, Dopamine agonist, Bile acid sequestrant, corticosteroids, methotrexate or immunosuppressive cytotoxic agents
* Some types of abdominal surgery, including bariatric surgery, or severe intestinal problems (by discretion of study physician), including:

  * Inflammatory bowel disease (IBD) including ulcerative colitis (mild-moderate-severe), Crohn s disease (mild-moderate-severe), or indeterminate colitis;
  * Irritable bowel syndrome (IBS) (moderate-severe);
  * Persistent, infectious gastroenteritis, colitis or gastritis, persistent or chronic diarrhea of unknown etiology, Clostridium difficile infection (recurrent) or Helicobacter pylori infection (untreated);
  * Chronic constipation
* Consumes more than 3 alcoholic beverages per day
* Currently receiving or has received antibiotics, antifungals, antivirals, or antiparasitics in past 2 months
* Is currently using or has used probiotic supplements within the last 2 months
* Is currently on a weight-loss program or has experienced a weight change (gain or loss) of greater than 15 pounds in the past 3 months
* Has a history of hospitalization for mental health condition and/or has had a change in depression or anxiety prescription medications within the past 10 weeks (by discretion of study physician)
* Is pregnant or breastfeeding or planning pregnancy within the time of the study
* Subjects who are not fluent in English
* Use of smoking or chewing tobacco, e-cigarettes, cigars, or other nicotine-containing products, or cannabis
* Regular use of prescription opiate pain medication
* Weight <100 lbs
* Acute disease, defined as the presence of a moderate or severe illness with or without fever, at the time of enrollment
* Inability to communicate effectively with study personnel
* Lack of commitment with the intervention or non-compliance (at the discretion of the investigator)
* Eating disorders

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2022-08-26 (Actual); Primary Completion 2026-02-04 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
The primary objective is to assess changes in gut microbiome associated with a Mediterranean-like and unprocessed food diet compared to a habitual Western diet in healthy adults. | 9 weeks (Short Term) 12 months (long Term)
  -Dietary intake via Dietary History Questionnaire (DHQ) III -PREDIMED MedDiet Score -Landry MedDiet Score -The CLEAN-MED NOVA score -Healthy Eating Index (HEI)-2015 -Weight change -Gut microbiome as measured by 16S rRNA analysis of frequent stool collections -Shotgun sequencing will include fungal and viral sequences -Microbial functional pathway analyses

SECONDARY OUTCOMES:
Measure biomarkers in various bodily specimens (stool, blood, etc.) using the pertinent biochemical assays. | 24 months
Identify associations between Mediterranean-like unprocessed food diet adherence with perceived quality of life. | 24 months
  -Daily assessment: CLEAN-MED Office for National Statistics (ONS) survey, 6 questions -Longer assessment: 36-Item Short Form Health Survey (SF-36) for health-related quality of life -Associations of changes in well-being with dietary patterns -Associations of changes in well-being with gut microbiota composition

CONTACTS AND LOCATIONS:
Overall Officials: David B Sacks, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
protocol was silent

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000871-CC.html